CLINICAL TRIAL: NCT01315392
Title: A Randomized Study of Immediate and Delayed Closure of Type II and IIIa Open Tibia Fractures: A Pilot Study
Brief Title: A Study of Immediate and Delayed Closure of Type II and IIIa Open Tibia Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Orthopaedic Trauma Association (Other); Orthopaedic Research and Education Fund (Unknown)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: OTAOREF2000MJB
Record Dates: First submitted 2011-03-01; First posted 2011-03-15 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2011-03

CONDITIONS: Type II and IIa Open Tibia Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- delayed closure (Active Comparator): wounds packed open with normal saline wet to dry gauze dressings and were returned to the operating room 36 to 72 hours after initial procedure for debridement and definitive closure.
  Interventions: Procedure: delayed closure
- immediate wound closure (Active Comparator): traumatic and surgical wounds closed at initial surgical intervention
  Interventions: Procedure: immediate wound closure

INTERVENTIONS:
Procedure: delayed closure — wounds packed open with normal saline wet to dry gauze dressings and were returned to the operating room 36 to 72 hours after initial procedure for a second debridement and definitive closure.
  Arms: delayed closure
Procedure: immediate wound closure — traumatic and surgical wounds closed at the initial surgical intervention
  Arms: immediate wound closure

SUMMARY:
Delayed wound closure is considered by many to be the standard of care for the treatment of an open fracture. This study was conducted to determine the feasibility of a large multi-center prospective randomized clinical trial and collect the pilot data needed to compete for the funding for such a trial. The study was designed to compare immediate and delayed closure of Gustilo type II and IIIa tibia diaphyseal fractures. The primary outcomes were the infection rates and fracture related complications in patients treated with immediate or delayed wound closure strategies.

ELIGIBILITY:
Inclusion Criteria:

* Gustilo type II-IIIa tibia fracture
* age greater than 15 years
* fractures amenable to intramedullary nailing

Exclusion Criteria:

* excessive wound contamination
* patient cardio-pulmonary or hemodynamic instability preventing prompt surgical intervention
* impaired or absent consciousness
* refusal of consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2000-07

PRIMARY OUTCOMES:
infection rate
  defined as cases determined definitively by a positive culture or treated empirically based on tenderness, erythema, and heat at the wound site.
hospital readmissions
  need for additional procedures and hospital readmissions related to the index injury will be documented
tibial fracture healing
  evidence of bridging callus on three of four cortices assessed by biplanar radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bosse, MD, Principal Investigator — Carolians HealthCare System
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States